CLINICAL TRIAL: NCT04069650
Title: Malnutrition is Not a Risk Factor for Free Flap Failure in the Oral Cavity
Acronym: FOOD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ZWETYENGA 2018
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Free Flap Reconstruction
MeSH Terms: interventions — Free Tissue Flaps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- None-malnutrition: normal nutritionnal status
  Interventions: Procedure: Free flap
- Malnutrition: * weight loss was superior to 5% in the past month;
  * a weight loss was superior to 10% in the past 6 months;
  * a BMI was inferior to 18,5 kg/m² (if age inferior to 70 years old) or inferior to 21 kg/m² (if age superior to > 70 years old) - a serum albumin level inferior to 30g/L (if age inferior to 70 years old) or inferior to <35g/L (if age superior to 70 years old).
  Interventions: Procedure: Free flap

INTERVENTIONS:
Procedure: Free flap — Free flap reconstruction of the oral cavity

SUMMARY:
Free flap reconstruction consists in replacing tissular defect from one body part by another tissu harvested in a distant site. Microsurgery has to be performed to restore vascularization.

Free flaps are now the gold standard in complex reconstruction. While reliable with a success rate superior to 95 %, a failure takes a heavy burden on the patient. Many risk factors have been highlitghted in free flap failure for head and neck microvascular reconstruction.

Among them, malnutrition is still debated. This is a retrospective cohort study comparing complications occurrence between two groups. One group with normal nutritionnal status, the other with malnutrition. Between january 2008 and january 2018, 70 patients who underwent oral cavity reconstruction using free flap were included. This is the first study known to date which uses clinical and biological variables to determine the nutritionnal status.

Malnutrition is not associated with a higher risk for free flap failure in the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* every consenting patients undergoing free flap reconstruction of the oral cavity

Exclusion Criteria:

* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing free flap reconstruction of the oral cavity
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Major complication occurency | 1 month
  in the first-month post-operative period, complications leading to flap loss

SECONDARY OUTCOMES:
Minor complication occurency | 1 month
  in the first-month post-operative period, complications NOT leading to flap loss

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France